CLINICAL TRIAL: NCT00003217
Title: A Pilot Study of Dose Intensification of Methotrexate and Cyclophosphamide in Patients With Advanced-Stage (III/IV) Small Non-Cleaved Non-Hodgkins Lymphoma and B-Cell All- A Limited Institution Phase III Pilot Study
Brief Title: Combination Chemotherapy in Treating Children With Stage III or Stage IV Non-Hodgkin's Lymphoma or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9517; POG-9517 (Other: Pediatric Oncology Group); CDR0000066078 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia; Lymphoma
Keywords: childhood Burkitt lymphoma; untreated childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; Doxorubicin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #26271; IND #7089
Drug: cytarabine
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #63878
Drug: dexamethasone
  Other Names: Decadron; NSC #034521
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127; IND #7038
Drug: methotrexate
  Other Names: MTX; amethopterin; NSC #740; IND #4291
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #67574; IND #7161

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy consisting of methotrexate and cyclophosphamide in treating children who have stage III or stage IV non-Hodgkin's lymphoma or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the feasibility and toxicity of dose intensification of methotrexate and cyclophosphamide in patients with stage III or IV small, noncleaved cell non-Hodgkin's lymphoma or B cell acute lymphoblastic leukemia. II. Estimate the response rate and survival of these patients after this therapy.

OUTLINE: This is a two-stage study. Patients will receive cytarabine either by continuous infusion (first stage) or bolus injection (second stage). Patients are stratified by disease (stage III non-Hodgkin's lymphoma (NHL) vs stage IV NHL vs stage B acute lymphoblastic leukemia). Therapy for all patients consists of alternating courses of "A" and "B". Patients with stage III disease receive 4 courses of chemotherapy (ABAB) while those with stage IV disease and B cell acute lymphoblastic leukemia receive 6 chemotherapy courses (ABABAB). Course A - Induction: Patients receive intrathecal methotrexate (IT MTX) and intrathecal cytarabine (IT Ara-C) on days 1, 4, and 11. Dexamethasone is administered by IV or orally twice a day on days 1-5. Cyclophosphamide IV is administered every 12 hours on days 1-3. Doxorubicin IV is administered over 15 minutes beginning 12 hours after the beginning of the 6th dose of cyclophosphamide (day 4). At the same time, vincristine IV is administered, then repeated on day 11. Patients begin filgrastim (granulocyte colony-stimulating factor; G-CSF) subcutaneously or IV over 30 minutes on day 5. Course B - Induction: The first 10 patients enrolled receive cytarabine by continuous infusion while the second 10 patients enrolled receive cytarabine by bolus IV. Patients begin treatment on day 18 and receive methotrexate IV over 24 hours plus IT MTX during hour 1. Dexamethasone is administered by IV or orally twice a day on days 1-5. After completing the 24 hour IV MTX infusion, patients begin cytarabine by continuous infusion over 48 hours or bolus IV every 12 hours for 4 doses. Patients receive G-CSF subcutaneously or IV over 30 minutes beginning on day 22. Patients are assessed for remission status before day 36. Course A - Consolidation: Patients receive dexamethasone IV or orally twice a day on days 1-5. IT MTX and IT Ara-C are administered on days 1 and 4. Cyclophosphamide is administered as during Induction, with vincristine IV and doxorubicin IV over 15 minutes 12 hours later. Vincristine repeats 1 week later. G-CSF administration begins on day 5. Course B - Consolidation: Therapy begins on day 22 with dexamethasone administered as previously. Methotrexate infusion and IT MTX are administered as in Course B - Induction, as is cytarabine (either as a continuous infusion or bolus IV). G-CSF is also administered as previously. Patients are followed monthly for the first 6 months, every 2 months for the next 6 months, then every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically proven small, noncleaved cell non-Hodgkin's lymphoma, Burkitt's lymphoma, non-Burkitt's lymphoma, or B cell acute lymphoblastic leukemia (B-ALL) Stage III or IV B-ALL - must have FAB L3 morphology and have been registered on POG-9400

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: HIV antibody positive allowed Not pregnant or lactating

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Prior emergency steroid therapy may be allowed Radiotherapy: Prior emergency radiotherapy may be allowed Surgery: Prior surgery allowed Other: No concurrent dexamethasone as an anti-emetic

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 1998-03; Primary Completion 2004-10 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C. Griffin, MD, Study Chair — Cook Children's Medical Center - Fort Worth
Locations (14):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Hospital for Sick Children, Toronto, Ontario